CLINICAL TRIAL: NCT02422121
Title: A Phase IIa Randomized, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Effects of Multiple Doses of Inhaled RNS60 and Budesonide on the Late Phase Asthmatic Response to Allergen Challenge in Patients With Mild Asthma. (This Study Has Been Amended to no Longer be a Cross Over Study; it Will be a Parallel (RNS60/Placebo) 1 Period Study and no Longer Involves the Administration of Budesonide)
Brief Title: Effect of RNS60 on the Late Phase Asthmatic Response to Allergen Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01.1.1.H3
Record Dates: First submitted 2015-04-14; First posted 2015-04-21 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — RNS60

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RNS60 (Experimental): RNS60, 4 ml twice daily
  Interventions: Drug: RNS60
- Placebo (Placebo Comparator): Normal Saline, 4 ml twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RNS60
  Arms: RNS60
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study will investigate the effect of treatment with RNS60 for 21 days. Subjects' FEV1 will be measured after an inhaled allergen challenge at baseline and again after 21 days of treatment.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, parallel study in approximately 32 male and female subjects with mild asthma. Each subject will receive either the experimental or the placebo, administered as a nebulized dose twice daily for 21 days.

ELIGIBILITY:
Inclusion Criteria

* Subjects who are able and willing to give written informed consent;
* Male and female subjects aged 18 to 65 years inclusive.
* Subjects with a body weight ≥50 kg and a BMI between 18.0 and 32.0 kg/m2 inclusive at screening.
* Subjects should be steroid-naïve (within 3 months of screening for oral corticosteroids and within 28 days of screening for inhaled corticosteroids) with mild asthma and satisfy the Global Initiative for Asthma (GINA) definition of asthma, but be otherwise healthy.
* Male subjects should agree to not donate sperm from first dose until 3 months post-last dose.
* Male subjects (with female partners of child bearing potential) and female subjects of child bearing potential should use two methods of highly effective contraception.
* Subjects should be non-smokers or ex-smokers for at least 12 months with less than a 10 pack year history.
* Subjects should not take any concomitant anti-asthma (except short-acting inhaled β2-agonists [SABAs]) or anti-allergy medication for at least 6 weeks prior to the screening visit and throughout the study period. Antihistamines will be permitted up to 7 days prior to the first screening visit.
* Pre-bronchodilator FEV1 of ≥70% of the predicted normal value for age, height and sex at screening and prior to first dose administration.
* Positive methacholine with a provocative concentration of methacholine resulting in a 20% fall in FEV1 (PC20 methacholine) of equal to or less than 8 mg/mL at screening.
* Documented allergy to at least one common allergen (house dust mite, grass pollen allergens or cat dander) as confirmed by a skin prick test wheal (≥3 mm in diameter). Historical data (up to 1 year) may be used.
* Early asthmatic response (FEV1 fall of ≥ 20%, 0 to 60 minutes after allergen challenge) and LAR (FEV1 fall of ≥15% 3 to 8 hours after challenge). Historical data up to 3 months before enrolment may be used.
* At admission FEV1 should be within 10% of the predicted FEV1 at screening. If subject does not meet this criterion at the first measurement 2 further repeats will be permitted.

Exclusion Criteria

* Subjects who do not conform to the above inclusion criteria.
* Female subjects who are pregnant, trying to become pregnant or lactating.
* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary (excluding mild asthma), gastrointestinal, cardiovascular (including ischemic heart disease), hepatic, psychiatric, neurologic, or severe allergies (e.g. anaphylaxis or angioedema).
* Worsening of asthma in the 4 weeks preceding the screening visit (requiring daily use of nebulised β2-agonists or any use of long acting β agonists [LABA], or requiring inpatient hospitalisation for asthma control, or requiring emergency room treatment, or requiring systemic corticosteroids for asthma control) or respiratory infection in the 4 weeks preceding the first screening visit or prior to randomization (Day 1).
* Use of any immunotherapy within 3 months prior to first screening.
* Use of nasal or inhaled corticosteroids, intraophthalmic corticosteroids, nasal, inhaled, or intraophthalmic cromolyn sodium or nedocromil, leukotriene receptor antagonists (zafirlukast, pranlukast, montelukast), and 5-lipoxygenase inhibitors (zileuton) within 28 days prior to first screening and throughout the study.
* Subject on LABA or short and long acting anti-muscarinics (SAMA or LAMA) see also Section 6.8.
* Concomitant disease or condition that could interfere with the conduct of the study, or for which the treatment could interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the patient in this study, including, but not limited to, cancer, alcoholism, drug dependency or abuse, or psychiatric disease.
* History of life-threatening asthma, defined as an asthma episode that required intubation or was associated with hypercapnoea, respiratory arrest or hypoxic seizures.
* Symptomatic with allergic rhinitis (e.g., hay fever), requiring treatment, at screening or predicted to have symptomatic allergic rhinitis (e.g., hay fever) during the time of study, requiring treatment.
* History of serious severe hypersensitivity or allergy (e.g., anaphylaxis).
* History of hypersensitivity to budesonide or to any of the excipients.
* Clinically significant abnormalities in physical examination or in laboratory test results (including serum biochemistry, hematology and urinalysis) as assessed by the Investigator.
* Subjects who have received any investigational drug in any clinical trial within 3 months, or who are on extended follow-up.
* Current diagnosis of active epilepsy or any active seizure disorder requiring chronic therapy with anti-epileptic drug(s).
* Subjects who are vegans or have medical dietary restrictions.
* Patients who take concomitant treatment with strong or moderate inhibitors of cytochrome P450 (CYP) 3A4 including oral/systemic ketoconazole, itraconozole, miconazole, clotrimazole, flucanazole, posaconazole, voriconazole, clarithromycin, erythromycin, ciprofloxacin, verapamil, diltiazem, indinavir, nelfinavir, saquinavir, ritonavir, amprenavir, lopinavir, atazanavir, darunavir and cyclosporine.
* Patients who take concomitant treatment with inducers of CYP3A4: carbamazepine, dexamethasone, phenytoin, rifabutin, rifampin and pioglitazone.
* Patients who take concomitant treatment with herbal medication/supplements or St John's Wort.
* Subjects with a supine systolic blood pressure ≥160 mmHg or a supine diastolic blood pressure ≥100 mmHg at screening or prior to randomization.
* History of alcohol abuse (intake of more than 24 units of alcohol per week) or drug addiction as seen on positive screen on drugs of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines) or positive alcohol test.
* Positive screen on hepatitis B surface antigen, antibodies to the hepatitis C virus or antibodies to the human immunodeficiency virus (HIV 1 and 2).
* Clinically significant abnormal 12-lead ECG or one demonstrating QTcB >450 ms at screening.
* Abnormal liver enzymes (alanine aminotransferase >1.5x upper limit of normal [ULN] or total bilirubin >1.5x ULN).
* Subjects who cannot communicate reliably with the Investigator.
* Subjects who are unlikely to co-operate with the requirements of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in late asthmatic response (LAR) as measured by spirometry | Baseline and Day 21
  The maximal percentage decrease from the pre-allergen challenge (post-diluent value) in FEV1 between 3 hours and 8 hours post-allergen challenge.

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Drug Research Unit at Guy's Hospital, London, United Kingdom